CLINICAL TRIAL: NCT05514444
Title: A Phase 1, Open-label, Multicenter Study of the Safety, Pharmacokinetics, and Pharmacodynamics of MK-4464 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced/Metastatic Solid Tumors
Brief Title: Study of MK-4464 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced/Metastatic Solid Tumors (MK-4464-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4464-001; MK-4464-001 (Other: MSD); 2023-504855-28-00 (Registry Identifier: EU CT); U1111-1290-2697 (Registry Identifier: UTN); 2021-005882-42 (EudraCT Number)
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Advanced/Metastatic Solid Tumors; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-4464 (Experimental): Participants will receive an intravenous (IV) infusion of MK-4464 administered in escalating doses every 3 weeks for up to 35 cycles. Escalation to subsequent MK-4464 doses will be based on safety of previous dose.
  Interventions: Biological: MK-4464
- MK-4464 + Pembrolizumab (Experimental): Participants will receive an IV infusion of MK-4464 administered in escalating doses and a 200 mg IV infusion of Pembrolizumab every 3 weeks for up to 35 cycles. Escalation to subsequent MK-4464 doses will be based on safety of MK-4464 monotherapy arm.
  Interventions: Biological: MK-4464; Biological: Pembrolizumab
- MK-4464 + Pembrolizumab + Zirconium 89 (89Zr)-MK-4464 (Experimental): Participants will receive an IV infusion of 89Zr-MK-4464 + IV infusion of MK-4464 on Cycle 1 Day 1, followed by an IV infusion of MK-4464 + a 200 mg IV infusion of pembrolizumab starting on Cycle 2 Day 1 and every 3 weeks for up to 35 cycles. Each cycle=3 weeks. MK-4464 doses will be based on safety of MK-4464 monotherapy arm. Participants may receive a 200 mg IV infusion of pembrolizumab on cycle 36.
  Interventions: Biological: MK-4464; Biological: Pembrolizumab; Drug: 89Zr-MK-4464

INTERVENTIONS:
Biological: MK-4464 — MK-4464 administered as an IV infusion every three weeks according to allocation and dose escalation.
Biological: Pembrolizumab — Pembrolizumab 200 mg administered as an IV infusion every three weeks.
  Arms: MK-4464 + Pembrolizumab; MK-4464 + Pembrolizumab + Zirconium 89 (89Zr)-MK-4464
Drug: 89Zr-MK-4464 — 89ZR-MK-4464 administered as an IV infusion on C1D1.
  Arms: MK-4464 + Pembrolizumab + Zirconium 89 (89Zr)-MK-4464

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics, and preliminary efficacy of MK-4464 as monotherapy and in combination with pembrolizumab in participants with advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

The key Inclusion Criteria include but are not limited to the following:

* Have a histologically or cytologically confirmed advanced/metastatic solid tumor by pathology report and have received, been intolerant to, been ineligible for, or refused all treatment known to confer clinical benefit
* Must submit a baseline tumor sample for analysis
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Human immunodeficiency virus (HIV) infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks, and have undetectable HBV viral load before randomization.

Exclusion Criteria:

The key Exclusion Criteria include but are not limited to the following:

* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) before the first dose of study intervention or has not recovered to CTCAE Grade 1 or better from any AEs that were due to cancer therapeutics administered more than 4 weeks earlier
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* Has clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active infection requiring therapy
* History of an allogenic stem cell transplant or a solid organ transplant
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has known psychiatric or substance abuse disorders that would interfere with the participant's ability to cooperate with the requirements of the study
* Has not fully recovered from any effects of major surgery without significant detectable infection
* Has received radiation therapy to the lung that is >30 gray (Gy) within 6 months of the first dose of study treatment
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Is currently participating and receiving study intervention in a study of an investigational agent or has participated and received study intervention in a study of an investigational agent or has used an investigational device within 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) | Up to approximately 21 days
  A DLT is any toxicity assessed by the investigator to be possibly, probably, or definitely related to study intervention administration that results in a change to a given dose or a delay in initiating the next cycle. All toxicities will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).
Number of Participants Who Experience At Least One adverse event (AE) | Up to approximately 27 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 24 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented.

SECONDARY OUTCOMES:
Minimum Plasma Concentration (Cmin) of MK-4464 | Once daily on Day 2, 3, 5, 8, 15 of Cycle 1 and 4, Pre-dose and immediately Post-dose Day 1 Cycle 1, 2, 3, 4, Pre-dose Day 1 Cycles 5, 6, 7, 8, and every 4 cycles thereafter through Cycle 35, 30 days post last dose (up to ~25 months); Cycle = 21 days
  Cmin is the minimum concentration of the drug observed in plasma. Blood samples will be collected pre-dose and post-dose at designated timepoints to determine Cmin of MK-4464.
Maximum Plasma Concentration (Cmax) of MK-4464 | Once daily on Day 2, 3, 5, 8, 15 of Cycle 1 and 4, Pre-dose and immediately Post-dose Day 1 Cycle 1, 2, 3, 4, Pre-dose Day 1 Cycles 5, 6, 7, 8, and every 4 cycles thereafter through Cycle 35, 30 days post last dose (up to ~25 months); Cycle = 21 days
  Cmax is the maximum concentration of the drug observed in plasma. Blood samples will be collected pre-dose and post-dose at designated timepoints to determine Cmax of MK-4464.
Area Under the Plasma Concentration-Time Curve (AUC) of MK-4464 | Once daily on Day 2, 3, 5, 8, 15 of Cycle 1 and 4, Pre-dose and immediately Post-dose Day 1 Cycle 1, 2, 3, 4, Pre-dose Day 1 Cycles 5, 6, 7, 8, and every 4 cycles thereafter through Cycle 35, 30 days post last dose (up to ~25 months); Cycle = 21 days
  AUC is a measure of the extrapolated mean concentration in serum. Blood samples will be collected pre-dose and post-dose at designated timepoints to determine AUC of MK-4464.
Objective Response Rate (ORR) | Up to 24 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by investigator assessment will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- The University of Louisville, James Graham Brown Cancer Center ( Site 0100), Louisville, Kentucky, United States
- Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0201), Toronto, Ontario, Canada
- Israel (2):
  - Rambam Health Care Campus-Oncology Division ( Site 0300), Haifa
  - Hadassah Medical Center-Oncology ( Site 0302), Jerusalem
- Netherlands (2):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek - NKI-AVL ( Site 0401), Amsterdam, North Holland
  - Amsterdam UMC, locatie VUmc ( Site 0400), Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26219&tenant=MT_MSD_9011